CLINICAL TRIAL: NCT03382730
Title: A Multi-centered Stepped Wedge Cluster Randomized Controlled Trial of the De-adoption of Oral Chlorhexidine Prophylaxis and Implementation of an Oral Care Bundle for Ventilated Critically Ill Patients
Brief Title: De-adoption of Oral Chlorhexidine Prophylaxis and Implementation of an Oral Care Bundle (CHORAL)
Acronym: CHORAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Toronto General Hospital (Other); University Health Network, Toronto (Other); Unity Health Toronto (Other); MOUNT SINAI HOSPITAL (Other)
Responsible Party: Principal Investigator, Craig M. Dale, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0913
Record Dates: First submitted 2017-10-19; First posted 2017-12-26 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Mortality; Oral Health; Dryness, Mouth; Pain, Orofacial
MeSH Terms: conditions — Xerostomia; Facial Pain | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Multi-centered stepped wedge cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Chlorhexidine Mouth Rinse (Other): Application of chlorhexidine gluconate mouth rinse per unit protocol.
  Interventions: Other: Chlorhexidine Mouth Rinse
- De-Adoption of Oral Chlorhexidine Mouth Rinse (Experimental): No application of chlorhexidine gluconate mouth rinse. Oral care bundle.
  Interventions: Other: Chlorhexidine Mouth Rinse De-Adoption

INTERVENTIONS:
Other: Chlorhexidine Mouth Rinse — Oral chlorhexidine gluconate oral rinse
  Other Names: Chlorhexidine
  Arms: Oral Chlorhexidine Mouth Rinse
Other: Chlorhexidine Mouth Rinse De-Adoption — Multifaceted education and audit/feedback.
  Other Names: De-adopt chlorhexidine
  Arms: De-Adoption of Oral Chlorhexidine Mouth Rinse

SUMMARY:
The objective of the CHORAL study is to evaluate the de-adoption of oral chlorhexidine and the introduction of a bundle of oral care practices on selected outcomes in critically ill mechanically ventilated adults.

DETAILED DESCRIPTION:
Infrequent or ineffective oral care can lead to mouth discomfort and lung infection for patients treated with ventilators (breathing machines) in intensive care units (ICUs). A commonly used mouthwash called chlorhexidine can reduce lung infection but most recent evidence shows it may increase the risk of death. In this study 6 participating intensive care units (ICUs) will de-adopt oral chlorhexidine and introduce a bundle of oral care practices using a multi-faceted educational tool kit. The investigators will measure changes in patient-oriented outcomes including mortality, ventilator-associated complications (VACs) and oral health status. A concurrent process evaluation will study how the intervention is delivered and received by patients and clinicians..

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive mechanical ventilation in the participating ICUs.

Exclusion Criteria:

* Does not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3260 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Intensive Care Unit (ICU) Mortality | 14 months
  All-cause mortality at time of ICU discharge

SECONDARY OUTCOMES:
Infection-related ventilator-associated complications (IVACs) | 14 months
  Changes in IVACs rates between groups
Beck Oral Assessment Score (BOAS), Modified | 14 months
  Changes in oral health between groups. Scores range from 5 (normal) to 20 (severe dysfunction).
Critical Care Pain Observational Tool (CPOT) | 14 months
  Changes in oropharyngeal pain between groups. CPOT scores range from 0-8 with a score >2 indicating presence of pain.
Oral Dryness - Numeric Rating Intensity Scale (NRS) | 14 months
  Changes in oral dryness scores between groups. NRS scores range from 0 (no dryness) to 10 (severe dryness).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Cuthbertson, MD FRCA, Principal Investigator — Sunnybrook Health Sciences Centre; Craig Dale, RN PhD, Principal Investigator — Sunnybrook Health Sciences Centre; University of Toronto
Locations (5):
- Canada (5):
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dale CM, Rose L, Carbone S, Smith OM, Burry L, Fan E, Amaral ACK, McCredie VA, Pinto R, Quinonez CR, Sutherland S, Scales DC, Cuthbertson BH. Protocol for a multi-centered, stepped wedge, cluster randomized controlled trial of the de-adoption of oral chlorhexidine prophylaxis and implementation of an oral care bundle for mechanically ventilated critically ill patients: the CHORAL study. Trials. 2019 Oct 24;20(1):603. doi: 10.1186/s13063-019-3673-0. PMID 31651364
- [Result] Dale CM, Rose L, Carbone S, Pinto R, Smith OM, Burry L, Fan E, Amaral ACK, McCredie VA, Scales DC, Cuthbertson BH. Effect of oral chlorhexidine de-adoption and implementation of an oral care bundle on mortality for mechanically ventilated patients in the intensive care unit (CHORAL): a multi-center stepped wedge cluster-randomized controlled trial. Intensive Care Med. 2021 Nov;47(11):1295-1302. doi: 10.1007/s00134-021-06475-2. Epub 2021 Oct 5. PMID 34609548